CLINICAL TRIAL: NCT06544928
Title: Utility of Remote Lung Auscultation in COPD With RESP™ Biosensor
Brief Title: Study on Home Obstructive Respiratory Exacerbations
Acronym: SHORE
Status: Enrolling by invitation | Type: Observational
Sponsor: Strados Labs, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SL-RS-SHORE
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: COPD Exacerbation; COPD (Chronic Obstructive Pulmonary Disease) With Acute Lower Respiratory Infection; COPD Exacerbation Acute; COPD
Keywords: SHORE; SL-RS-SHORE; RESP™ Biosensor; RESP™; Strados Labs
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All Subjects: Device: RESP Biosensor The RESP Biosensor will be placed on all qualitfying subjects for recording of auscultory sound.
  Interventions: Device: RESP™ Biosensor

INTERVENTIONS:
Device: RESP™ Biosensor — For this observational study, the RESP™ Biosensor will be placed on the patient for periodic recording of auscultory sound.

SUMMARY:
Strados Labs has developed the Strados™ Respiratory Care Platform, including the RESP™ Biosensor System, which encompasses a clinically validated wearable, non-invasive, Bluetooth-enabled device capable of remotely collecting respiratory data. RESP was designed to extend both the geographical and temporal range of lung sound recordings, which can improve the remote monitoring of high-risk COPD patients. The RESP Biosensor continuously captures lung sounds and chest wall motions that are wirelessly transmitted through a mobile app to a web application to be analyzed for changes in respiratory health.

Preliminary data suggest good patient compliance and the potential for RESP to detect early COPD exacerbation. However, uncertainty on the optimal RESP monitoring procedure and insufficient longitudinal RESP data for definitive statistical correlation with COPD exacerbations warrant further study.

We plan to conduct an observational study to assess feasibility of home RESP remote patient monitoring and secondarily collect the longitudinal data necessary to establish the correlation between RESP based measures and standard of care measures of COPD symptom severity.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 40 and 80 with documented physician-diagnosed COPD and FEV1/FVC<0.70 or LLN based on post-bronchodilator spirometry

* Hospitalized for COPD exacerbation with plan for discharge within 48 hours OR
* Visiting pulmonologist post COPD-exacerbation within 14 days of discharge from hospital 3. Tobacco History: Current or Former Smoker
* Has smoked at least 100 cigarettes in his/her lifetime 4. Patient can follow study procedures, including instructions for self-placement and operation of biosensor
* Patient has experience/owns a smartphone 5. Patient is accessible by telehealth/telephone for duration of the study 6. Patient is able and willing to return to study site for study visits as necessary

Exclusion Criteria:

1. Patient is unable or unwilling to provide informed consent
2. Any condition that, in the opinion of the investigator, would limit the patient's activity in the study and/or adequate lung sound capture using the RESP™ wearable device
3. Patient with end-stage medical condition with expected survival no more than 6 months
4. History of adverse reaction or allergy to adhesives such as TegaDerm®

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are hospitalized for COPD exacerbation with plan for discharge within 48 hoursare, OR are visiting their pulmonologist in the outpatient setting or via telehealth within 14 days of a COPD exacerbation with inpatient stay.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
The study will assess observational outcome measures. No formal efficacy or safety endpoints are defined. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jefferson Einstein Philadelphia Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided